CLINICAL TRIAL: NCT06345560
Title: Pharmacokinetics of Drospirenone Only Pills in Obese Thai Women: A Pre- and Post-Bariatric Surgery Study
Brief Title: Pharmacokinetics of Drospirenone Only Pills: A Pre- and Post-Bariatric Surgery Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 077766
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-03

CONDITIONS: Contraception
Keywords: Drospirenone only pills; Obesity; Bariatric surgery; Roux-en-Y gastric bypass; Pharmacokinetics; Absorption
MeSH Terms: conditions — Obesity | interventions — drospirenone

STUDY DESIGN:
Intervention Model Description: Pre-bariatric surgery pharmacokinetics study of Drospirenone compare with post-bariatric surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Drospirenone (Experimental): Participants received Drospirenone 4 mg tablet orally once daily for 21-28 days
  Interventions: Drug: Drospirenone

INTERVENTIONS:
Drug: Drospirenone — 4 mg tablet once daily

SUMMARY:
The purpose of this study is to investigate whether bariatric surgery affects Drospirenone only pills absorption

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants giving written informed consent who meet the eligibility requirements will take Drospirenone-only pills (4 mg, once daily). Between the 21st and 28th day of Drospirenone taking, pharmacokinetics will be measured. Pre-bariatric surgery pharmacokinetics study will be compared with post-bariatric surgery pharmacokinetics study.

ELIGIBILITY:
Inclusion Criteria:

* Thai women aged 18-45 years who are obese and had an appointment for Bariatric surgery at Chulalongkorn Hospital
* Need contraception
* Able to use non-hormonal contraception during the study
* Giving consent

Exclusion Criteria:

* Pregnancy or history of giving birth within 3 months
* Breastfeeding within the 6 months
* History of using DMPA within 12 months
* History of using other types of hormonal birth control pills within 4 weeks
* History of bilateral oophorectomy or hysterectomy
* Suspected ovarian tumor or pathological ovarian cyst
* Regular cigarette smoking
* Contraindications to Drospirenone

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration versus Time of Drospirenone | 1 month before and 1 month after bariatric surgery
  Plasma concentration of Drospirenone will be measured at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8 hours post-dose

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Punyawee Utaipatanacheep, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Currently have no recruited participants. You can ask for information directly from the investigators in future.

REFERENCES:
- [Result] Techagumpuch A, Pantanakul S, Chansaenroj P, Boonyagard N, Wittayapairoch J, Poonthananiwatkul T, et al. Thai Society for metabolic and bariatric surgery consensus guideline on bariatric surgery for the treatment of obese patient in Thailand. JAGST 2021;4:5-18.
- [Result] Simmons K, Edelman A. Contraception in the setting of obesity and bariatric surgery. In: Allen RH, Cwiak CA, editors. Contraception for the medically challenging patient. New York: Springer; 2014. P. 157-80.
- [Result] ACOG practice bulletin no. 105: bariatric surgery and pregnancy. Obstet Gynecol. 2009 Jun;113(6):1405-1413. doi: 10.1097/AOG.0b013e3181ac0544. No abstract available. PMID 19461456
- [Result] Ciangura C, Coupaye M, Deruelle P, Gascoin G, Calabrese D, Cosson E, Ducarme G, Gaborit B, Lelievre B, Mandelbrot L, Petrucciani N, Quilliot D, Ritz P, Robin G, Salle A, Gugenheim J, Nizard J; BARIA-MAT Group. Clinical Practice Guidelines for Childbearing Female Candidates for Bariatric Surgery, Pregnancy, and Post-partum Management After Bariatric Surgery. Obes Surg. 2019 Nov;29(11):3722-3734. doi: 10.1007/s11695-019-04093-y. PMID 31493139
- [Result] Mechanick JI, Apovian C, Brethauer S, Timothy Garvey W, Joffe AM, Kim J, Kushner RF, Lindquist R, Pessah-Pollack R, Seger J, Urman RD, Adams S, Cleek JB, Correa R, Figaro MK, Flanders K, Grams J, Hurley DL, Kothari S, Seger MV, Still CD. Clinical Practice Guidelines for the Perioperative Nutrition, Metabolic, and Nonsurgical Support of Patients Undergoing Bariatric Procedures - 2019 Update: Cosponsored by American Association of Clinical Endocrinologists/American College of Endocrinology, The Obesity Society, American Society for Metabolic and Bariatric Surgery, Obesity Medicine Association, and American Society of Anesthesiologists. Obesity (Silver Spring). 2020 Apr;28(4):O1-O58. doi: 10.1002/oby.22719. PMID 32202076
- [Result] Mengesha BM, Carter JT, Dehlendorf CE, Rodriguez AJ, Steinauer JE. Perioperative pregnancy interval, contraceptive counseling experiences, and contraceptive use in women undergoing bariatric surgery. Am J Obstet Gynecol. 2018 Jul;219(1):81.e1-81.e9. doi: 10.1016/j.ajog.2018.04.008. Epub 2018 Apr 7. PMID 29634911
- [Result] United Nations Department of Economic and Social Affairs, Population Division (2022). World Contraceptive Use 2022 [Internet]. [cited 9 August 2023]. Available from: https://www.un.org/development/desa/pd/data/world-contraceptive-use.
- [Result] Nightingale AL, Lawrenson RA, Simpson EL, Williams TJ, MacRae KD, Farmer RD. The effects of age, body mass index, smoking and general health on the risk of venous thromboembolism in users of combined oral contraceptives. Eur J Contracept Reprod Health Care. 2000 Dec;5(4):265-74. doi: 10.1080/13625180008500402. PMID 11245554
- [Result] Jick H, Jick SS, Gurewich V, Myers MW, Vasilakis C. Risk of idiopathic cardiovascular death and nonfatal venous thromboembolism in women using oral contraceptives with differing progestagen components. Lancet. 1995 Dec 16;346(8990):1589-93. doi: 10.1016/s0140-6736(95)91928-7. PMID 7500750
- [Result] Effect of different progestagens in low oestrogen oral contraceptives on venous thromboembolic disease. World Health Organization Collaborative Study of Cardiovascular Disease and Steroid Hormone Contraception. Lancet. 1995 Dec 16;346(8990):1582-8. PMID 7500749
- [Result] Rosano GMC, Rodriguez-Martinez MA, Spoletini I, Regidor PA. Obesity and contraceptive use: impact on cardiovascular risk. ESC Heart Fail. 2022 Dec;9(6):3761-3767. doi: 10.1002/ehf2.14104. Epub 2022 Sep 14. PMID 36103980
- [Result] Cardiovascular disease and use of oral and injectable progestogen-only contraceptives and combined injectable contraceptives. Results of an international, multicenter, case-control study. World Health Organization Collaborative Study of Cardiovascular Disease and Steroid Hormone Contraception. Contraception. 1998 May;57(5):315-24. PMID 9673838
- [Result] Vasilakis C, Jick H, del Mar Melero-Montes M. Risk of idiopathic venous thromboembolism in users of progestagens alone. Lancet. 1999 Nov 6;354(9190):1610-1. doi: 10.1016/S0140-6736(99)04394-9. PMID 10560680
- [Result] WHO Guidelines Approved by the Guidelines Review Committee. Medical Eligibility Criteria for Contraceptive Use. 5 ed. Geneva: World Health Organization Copyright © World Health Organization 2015.; 2015. p. 156-85.
- [Result] Curtis KM, Tepper NK, Jatlaoui TC, Berry-Bibee E, Horton LG, Zapata LB, Simmons KB, Pagano HP, Jamieson DJ, Whiteman MK. U.S. Medical Eligibility Criteria for Contraceptive Use, 2016. MMWR Recomm Rep. 2016 Jul 29;65(3):1-103. doi: 10.15585/mmwr.rr6503a1. PMID 27467196
- [Result] Palacios S, Colli E, Regidor PA. Efficacy and cardiovascular safety of the new estrogen-free contraceptive pill containing 4 mg drospirenone alone in a 24/4 regime. BMC Womens Health. 2020 Oct 2;20(1):218. doi: 10.1186/s12905-020-01080-9. PMID 33008401
- [Result] Palacios S, Regidor PA, Colli E, Skouby SO, Apter D, Roemer T, Egarter C, Nappi RE, Skrivanek A, Jakimiuk AJ, Weyers S, Acs N, Elia D, Gemzell Danielsson K, Bitzer J. Oestrogen-free oral contraception with a 4 mg drospirenone-only pill: new data and a review of the literature. Eur J Contracept Reprod Health Care. 2020 Jun;25(3):221-227. doi: 10.1080/13625187.2020.1743828. Epub 2020 Apr 21. PMID 32312141
- [Result] Creinin MD, Angulo A, Colli E, Archer DF. The efficacy, safety, and tolerability of an estrogen-free oral contraceptive drospirenone 4 mg (24/4-day regimen) in obese users. Contraception. 2023 Dec;128:110136. doi: 10.1016/j.contraception.2023.110136. Epub 2023 Aug 5. PMID 37544572
- [Result] Archer DF, Ahrendt HJ, Drouin D. Drospirenone-only oral contraceptive: results from a multicenter noncomparative trial of efficacy, safety and tolerability. Contraception. 2015 Nov;92(5):439-44. doi: 10.1016/j.contraception.2015.07.014. Epub 2015 Jul 29. PMID 26232513
- [Result] Schlatter J. Oral Contraceptives after Bariatric Surgery. Obes Facts. 2017;10(2):118-126. doi: 10.1159/000449508. Epub 2017 Apr 22. PMID 28433989
- [Result] Andersen AN, Lebech PE, Sorensen TI, Borggaard B. Sex hormone levels and intestinal absorption of estradiol and D-norgestrel in women following bypass surgery for morbid obesity. Int J Obes. 1982;6(1):91-6. PMID 7068318
- [Result] Victor A, Odlind V, Kral JG. Oral contraceptive absorption and sex hormone binding globulins in obese women: effects of jejunoileal bypass. Gastroenterol Clin North Am. 1987 Sep;16(3):483-91. PMID 2449395
- [Result] Weiss HG, Nehoda H, Labeck B, Hourmont K, Marth C, Aigner F. Pregnancies after adjustable gastric banding. Obes Surg. 2001 Jun;11(3):303-6. doi: 10.1381/096089201321336647. PMID 11433905
- [Result] Gerrits EG, Ceulemans R, van Hee R, Hendrickx L, Totte E. Contraceptive treatment after biliopancreatic diversion needs consensus. Obes Surg. 2003 Jun;13(3):378-82. doi: 10.1381/096089203765887697. PMID 12841897
- [Result] Ginstman C, Frisk J, Carlsson B, Arlemalm A, Hagg S, Brynhildsen J. Plasma concentrations of etonogestrel in women using oral desogestrel before and after Roux-en-Y gastric bypass surgery: a pharmacokinetic study. BJOG. 2019 Mar;126(4):486-492. doi: 10.1111/1471-0528.15511. Epub 2018 Nov 16. PMID 30347490
- [Result] Moreira de Brito C, de Melo ME, Mancini MC, Santo MA, Cercato C. Pharmacokinetics of oral levonorgestrel and ethinylestradiol in women after Roux-en-Y gastric bypass surgery. Surg Obes Relat Dis. 2021 Apr;17(4):673-681. doi: 10.1016/j.soard.2020.12.007. Epub 2020 Dec 16. PMID 33547015
- [Result] UK Medical Eligibility Criteria For Contraceptive Use UKMEC 2016 (amended September 2019). UK: the Faculty of Sexual and Reproductive Healthcare; 2019.
- [Result] FSRH Guideline (August 2022) Progestogen-only Pills. BMJ Sex Reprod Health. 2022 Aug;48(Suppl 1):1-75. doi: 10.1136/bmjsrh-2022-PoP. No abstract available. PMID 36316023
- [Result] Richter WH, Koytchev R, Kirkov V, Merki G, Colli E, Regidor PA. Comparative pharmacokinetic estimates of drospirenone alone and in combination with ethinyl estradiol after single and repeated oral administration in healthy females. Contraception. 2020 Feb;101(2):137-143. doi: 10.1016/j.contraception.2019.10.005. Epub 2019 Nov 21. PMID 31758920
- [Result] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848